CLINICAL TRIAL: NCT04150016
Title: Assessment of In-stent Intimal Repair and Vessel Reaction After FirehawkTM Sirolimus Eluting Stent Implantation of STEMI Subjects - An Optical Coherence Tomography (OCT) Study
Brief Title: In-stent Repair and Vessel Reaction of STEMI Patients With OCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XijingH-OCT
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Drug-eluting Stents; Percutaneous Coronary Intervention; Optical Coherence Tomography; ST-Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Firehawk implantation (Experimental): 22 subjects will be enrolled to receive Firehawk™ sirolimus target-eluting stent(s).
  Interventions: Procedure: percutaneous coronary intervention
- XIENCE implantation (Active Comparator): 22 subjects will be enrolled to receive XIENCE™ everolimus target-eluting stent(s).
  Interventions: Procedure: percutaneous coronary intervention

INTERVENTIONS:
Procedure: percutaneous coronary intervention — Percutaneous coronary intervention (PCI), also known as coronary angioplasty, is a nonsurgical procedure that improves blood flow to your heart.PCI requires cardiac catheterization, which is the insertion of a catheter tube and injection of contrast dye, usually iodine-based, into your coronary arteries. Doctors use PCI to open coronary arteries that are narrowed or blocked by the buildup of atherosclerotic plaque. PCI may be used to relieve symptoms of coronary heart disease or to reduce heart damage during or after a heart attack.
  Other Names: PCI

SUMMARY:
This study is a prospective, multi-center, non-inferior, randomized controlled clinical trial, aims to use optical Coherence tomography to observe the the early- and mid-stage vessel repair and neointimal proliferation. And to assess the safety and effectiveness of the Firehawk™ sirolimus target-eluting coronary stent system with abluminal grooves containing a biodegradable polymer (Firehawk™) comparing the XIENCE everolimus-eluting coronary stent system in the treatment of subjects with ST-elevation myocardial infarction (STEMI).

ELIGIBILITY:
Clinical Inclusion Criteria:

CI1. Subject must be 18 - 75 years of age; male or female without pregnancy.

CI2. Subjects recently suffer from SETMI (from 20 minute to 12 hours), and ECG changes consistent with AMI:

* 1mm elevation in more than 2 continuously leads, or; Newly developed LBBB, or;
* 1mm depression in more than 2 continuously leads representing Posterior myocardial infarction) CI3. New, in situ and single or bifurcation lesion of target vessel. CI4. Subject only implanted one brand of stent. CI5. Subjects are eligible candidates for coronary artery bypass graft surgery (CABG).

CI6. Subject (or legal guardian) understands the trial requirements and the treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed;

Angiographic Inclusion Criteria:

AI1. At least one of the target lesions must be acute occlusion lesion, and Eligible for percutaneous coronary intervention (PCI), and Having a visually estimated diameter restenosis no less than 70% (or a visually estimated diameter restenosis no less than 50% with consistent clinical symptoms), TIMI blood flow no less than Grade I, and have a visually estimated reference diameter ≥2.25 mm and ≤4.0 mm.

AI2. Target lesions must be able to pass through all target lesions (no severe tortuosity or calcification in proximal lesion).

AI3. Target lesions of type A lesion defined by ACC/AHA must be successfully expanded (no severe calcification in target lesion).

Clinical Exclusion Criteria:

CE1. Subjects with Cardiogenic shock. CE2. Subjects with severe heart failure (NYHA classification ≥ 3) or LVEF<35%. CE3. Subjects with elevated serum creatinine level >2.0mg/dL or undergoing dialysis therapy.

CE4. Subjects associated with drugs allergy (such as sirolimus, everolimus, stent alloys, contrast medium, heparin, clopidogrel or aspirin).

CE5. Subjects with bleeding tendency, active peptic ulcer, active gastrointestinal (GI) bleeding or other bleeding diathesis or coagulopathy, or refused a blood transfusion.

CE6. Subjects with cardiac stroke or with sequelae of stroke. CE7. Subjects with cebral tumor, Cerebral aneurysms, cerebral arteriovenous malformation (AVM), transient ischemic attack (TIA), permanent nerve defects, GI bleeding within 2 months, major operation within 6 weeks, or with abnormal counts of platelet and hemoglobin (Hb): platelet counts less than 1×106/mm3, Hb less than 10g/dL.

CE8. Subjects plan to undergo any operations within 6 months that may lead to anti-platelet therapy discontinuation.

CE9. Subjects are suffering from other serious illness, which may cause drop in life expectancy to less than 12 months.

CE10. Subjects were participating in another study of drug or medical device, which did not meet its primary endpoint.

CE11. Subject are considered unwilling to understand the trial requirements and refused to follow the treatment procedures.

CE12. Subject with Heart transplantation.

Angiographic Exclusion Criteria:

AE1. Target lesions with true bifurcation lesion (both main and branch vessel need implantation).

AE2. Target lesions with unprotected left main. AE3. Target lesions with more than 100mm in length. AE4. Target lesions with in-stent stenosis. AE5. Uncertain target lesions. AE6. Target lesion unsuitable for 6 months OCT follow up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2019-03-08 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Neointimal thickness by OCT | At 6 months post-index procedure

SECONDARY OUTCOMES:
Percentage of Uncovered Struts by OCT | At 6 months post-index procedure
Target lesion failure | 30 days, 6 months, 12 months post-index procedure
Percentage of Malaposition Struts by OCT | At 6 months post-index procedure
Thrombosis (from ARC definition) | 30 days, 6 months, 12 months post-index procedure
In-stent and in-segment late lumen loss | At 6 months post-index procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] He Y, Wang R, Liu J, Li F, Li J, Li C, Zhou J, Zhao Z, Yang W, Mou F, Wang J, Kan J, Li X, Li Y, Zheng M, Chen S, Gao C, Tao L. A Randomized Comparison of the Healing Response Between the Firehawk Stent and the Xience Stent in Patients With ST-Segment Elevation Myocardial Infarction at 6 Months of Follow-Up (TARGET STEMI OCT China Trial): An Optical Coherence Tomography Study. Front Cardiovasc Med. 2022 Jun 1;9:895167. doi: 10.3389/fcvm.2022.895167. eCollection 2022. PMID 35722108